CLINICAL TRIAL: NCT06604689
Title: Artificial Intelligence-guided Prognostication and Cranial Radiotherapy Optimization in First-line Third-generation EGFR-TKI-treated EGFR-mutant Non-small Cell Lung Cancer With Baseline Brain Metastases: a Multicenter, Observational Study
Brief Title: AI-guided Prognostication and Cranial Radiotherapy Optimization in EGFR-TKI-treated Non-small Cell Lung Cancer Patients With Baseline Brain Metastases
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Other Study IDs: BM-AI
Record Dates: First submitted 2024-09-18; First posted 2024-09-19 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); Brain Metastasases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Construction of AI models (retrospective cohort)
  Interventions: Drug: third-generation EGFR TKIs (Almonertinib/Furmonertinib/Osimertinib)
- Validation of AI models (prospective cohort)
  Interventions: Drug: third-generation EGFR TKIs (Almonertinib/Furmonertinib/Osimertinib)

INTERVENTIONS:
Drug: third-generation EGFR TKIs (Almonertinib/Furmonertinib/Osimertinib) — EGFR-mutated NSCLC patients with brain metastases who met the inclusion and exclusion criteria, would receive first-line third-generation EGFR-TKI treatment (monotherapy or combined with upfront cranial radiotherapy)

SUMMARY:
The goal of this observational study is to extract the imaging features of brain lesions and primary lung lesions in NSCLC patients with brain metastases by deep learning, as well as common clinicopathological parameters, which are used to construct a multimode model that can accurately predict the treatment efficacy and survival of the third-generation EGFR-TKI treatment, and to use the model to assist in screening high-risk populations suitable for upfront cranial radiotherapy.

Participants receiving third-generation EGFR-TKI treatment will be enrolled in our study and we will collect their regular contrast-enhanced chest CT and contrast-enhanced brain MRI for model construction.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non-small cell lung cancer;
* clinical stage IV (AJCC, 8th edition, 2017);
* EGFR sensitive mutations: EGFR L858R, EGFR exon 19 deletion;
* age≥18 years old;
* KPS score≥70;
* brain metastases at diagnosis;
* complete systemic imaging (including brain MRI) before third-generation EGFR-TKI treatment;
* received standard third-generation EGFR-TKI therapy (monotherapy or combined with brain radiotherapy);
* willing to cooperate with the follow-up after third-generation EGFR-TKI treatment;
* informed consent of the patient.

Exclusion Criteria:

* Multiple primary or metastatic tumors (except early skin cancer, cervical carcinoma in situ that has been treated radically, with no recurrence or progression for more than 5 years);
* Pregnant or lactating women who, as judged by the investigator, were not candidates for brain MRI;
* EGFR sensitive mutations were negative or EGFR mutation status was not detected.
* Uncontrolled epilepsy, central nervous system disease, or history of mental disorders, judged by the researcher to potentially interfere with the signing of the informed consent form or affect patient compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are collected all over china, diagnosed with EGFR-mutant NSCLC with brain metastases.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 1 year
  The time from the start of EGFR-TKI treatment until the documentation of disease progression or death from any cause, assessed according to the RECIST 1.1 criteria. Patients who are still alive at the time of analysis will have their last contact date used as the cutoff date.

SECONDARY OUTCOMES:
Intracranial Objective Response Rate (iORR) | 1 year
  The percentage of participants in the analysis population whose brain lesions achieve CR or PR, assessed according to the modified RECIST 1.1 criteria.
Intracranial Progression-Free Survival (iPFS) | 1 year
  The time from the start of EGFR-TKI treatment until the documentation of intracranial disease progression or death from any cause. If the patients have extracranial disease progression (without intracranial disease progression), the cutoff date was the date of the first occurrence of extracranial disease progression. Patients who have not progressed at the time of analysis will have their last contact date used as the cutoff date.
Overall Survival (OS) | 1 year
  The time from the start of EGFR-TKI treatment until death from any cause. Patients who are still alive at the time of analysis will have their last contact date used as the cutoff date.
Objective Response Rate (ORR) | 1 year
  The percentage of participants who achieve a Complete Response (CR) or Partial Response (PR) after treatment, assessed according to the RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer center, Shanghai, Shanghai Municipality, China